CLINICAL TRIAL: NCT04885673
Title: High Flow Nasal Cannula in Comparison to Apneic Oxygenation During Foreign Body Removal by Rigid Bronchoscope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, samar mohammed, Lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FMASU R101/2021
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (High flow nasal cannula group) (Active Comparator): (Vapotherm) will be used during the bronchoscopy time flow rate 50 L/min with 100% humidified oxygen and the temperature adjusted to be 38℃
  Interventions: Device: Vapotherm
- Group B (Apeieoc oxygenation group) (Active Comparator): The standard apneic oxygenation through the side port of rigid bronchoscope during the procedure
  Interventions: Device: Apneic oxygenation

INTERVENTIONS:
Device: Vapotherm — flow rate 50 L/min with 100% humidified oxygen and the temperature adjusted to be 38℃
  Other Names: High flow nasal cannula
  Arms: Group A (High flow nasal cannula group)
Device: Apneic oxygenation — Standard apneic oxygenation through the side port of rigid bronchoscope during the procedure
  Arms: Group B (Apeieoc oxygenation group)

SUMMARY:
To compare the effect of HFNC with standard apneic oxygenation on patient oxygenation and airway protection during foreign body removal by rigid bronchoscope.

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled trial, at Ain Shams University hospitals, Cardiovascular surgery hospital (Thoracic surgery unit), Cairo, Egypt. We will include 64 patients planned for foreign body removal by rigid bronchoscope. All patients will be ASA І with recent FB aspiration in the last 72hrs either by history or documented by radiopaque shadow in chest X ray or CT scan. After achievement of anesthesia and full muscle relaxation ventilation started by open mask technique. Then the patients will be divided into two groups according to the oxygenation technique:

Group (A) (32 patients) HFNC (Vapotherm) will be used during the bronchoscopy time flow rate 50 L/min with 100% humidified oxygen and the temperature adjusted to be 38℃ .

Group (B) (32 patients) (control group) using the standard apneic oxygenation through the side port of rigid bronchoscope during the procedure

ELIGIBILITY:
Inclusion Criteria:

* We will include 64 patients planned for foreign body removal by rigid bronchoscope.
* All patients will be ASA І
* Recent FB aspiration in the last 72hrs either by history or documented by radiopaque shadow in chest X ray or CT scan.

Exclusion Criteria:

* Patients age not more than 40 years old.
* Body weight less than 40 kg.
* Critically ill patients.
* Intubated patients.
* Inhalation of FB more than 72 hrs.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-04-25 (Actual); Primary Completion 2021-07-05 (Estimated); Study Completion 2021-07-25 (Estimated)

PRIMARY OUTCOMES:
Maintain high level of oxygen saturation during the procedure | During the procedure time
  Monitoring oxygen saturation by pulse oximeter and recording the readings

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Mohammed, Cairo, Egypt